CLINICAL TRIAL: NCT04691570
Title: A Phase 2, Open-Label, Repeat Dose Study to Assess the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of Intravenous ANX005 in Subjects With Warm Autoimmune Hemolytic Anemia (wAIHA)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ANX005 in Participants With Warm Autoimmune Hemolytic Anemia (wAIHA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANX005-wAIHA-02
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Warm Autoimmune Hemolytic Anemia (wAIHA)
Keywords: AIHA; C1q; complement; RBC lysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ANX005 (Experimental): Participants will receive two once-weekly doses of ANX005 at specific time points
  Interventions: Drug: ANX005

INTERVENTIONS:
Drug: ANX005 — ANX005 is provided as a solution for IV infusion

SUMMARY:
This study will evaluate the safety and tolerability of ANX005 in participants with Warm Autoimmune Hemolytic Anemia (wAIHA).

DETAILED DESCRIPTION:
After being informed of study details and potential risks, all participants who provide written informed consent will undergo an up to 6-week screening period to determine eligibility. Participants who meet the eligibility criteria will receive two once-weekly intravenous (IV) infusions of ANX005. Participants will return to the clinic weekly through Week 10 for study assessments. The total duration of individual participation in this study will be up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female ≥18 years of age (no maximum age).
* Diagnosis of wAIHA at least 3 months prior to screening with a direct antiglobulin test (DAT) ≥1 positive for immunoglobulin G (IgG)±C3, or a diagnosis of mixed autoimmune hemolytic anemia (AIHA) that is DAT positive for both IgG and C3, with a presence of a cold antibody with a thermal amplitude ≥30ºCelcius.
* Hemoglobin (Hgb) level ≤10.0 grams/deciliter (pre-transfusion).
* Evidence of classical complement pathway activation.
* Evidence of active hemolysis.
* Stable use of glucocorticoids and immunosuppressants are permitted.
* Vaccinations against encapsulated bacterial organisms within 5 years prior to screening or participant must be willing to receive prophylaxis against infections with encapsulated bacteria via vaccination and/or the use of prophylactic antibiotics in accordance with local standards of practice and/or guidelines.

Exclusion Criteria:

* Elevated aspartate aminotransferase or alanine aminotransferase levels >2.5 times the upper limit of normal.
* Platelet count <30 X 10^9/liter.
* History of cold agglutinin disease.
* History of solid organ, bone marrow, or stem cell transplantation.
* History of splenectomy within the 3 months prior to screening.
* Received rituximab or other anti-CD20 monoclonal antibody <3 months prior to screening.
* Intravenous immunoglobulin (IVIg) treatment within 3 months prior to screening or plasmapheresis or immunoadsorption treatment within 60 days prior to screening.
* Clinically significant, recent, or ongoing illness or medical condition, including coexistent autoimmune disorder, malignancy, HIV, hepatitis B virus, and hepatitis C virus.
* History of meningitis or septicemia within the past 2 years.
* Treatment with an investigational therapeutic agent within 30 days prior to screening.
* Hypersensitivity to any drug product or excipients used in this study or to previous IV medication administration.
* Body weight less than 50 kilograms (kg) or greater than 100 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Safety: Treatment-emergent adverse events (TEAEs) | Up to Week 16
  Number of participants with TEAEs, defined as any adverse event with an onset on or after the day of infusion through 16 weeks after the infusion
Change in disease activity biomarkers | Baseline to Day 71
  Change in hemoglobin, lactate dehydrogenase, bilirubin, reticulocyte count and haptoglobin from baseline

SECONDARY OUTCOMES:
Plasma concentrations | Up to Day 71
  Plasma concentrations of ANX005 over time
Change in complement system biomarkers | Baseline to Day 71
  Change in CH50 and C1q from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Annexon, Inc.
Locations (1):
- Investigational Site 01, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No